CLINICAL TRIAL: NCT07146113
Title: A Multicentre Observational Study on Treatment Approaches and Biomarkers in de Novo Metastatic Hormone Sensitive Prostate Cancer in Russian Federation
Brief Title: Treatment Approaches and Biomarkers PRevalence In de Novo MEtastatic Hormone-sensitive Prostate Cancer in Russian Federation
Acronym: PRIME
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133HR00058
Record Dates: First submitted 2025-06-26; First posted 2025-08-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
A multicentre observational study on treatment approaches and biomarkers in de novo metastatic hormone sensitive prostate cancer in Russian Federation

DETAILED DESCRIPTION:
This is a multicentre observational study on treatment approaches, demographic and clinical characteristics and prevalence of biomarkers (PTEN-loss, HER2-positive status; HRR mutations, HRD-positive status) in patients with de novo high-aggressive mHSPC in Russian Federation. The study will sequentially include only those patients who have signed the informed consent form (ICF). No procedures will be applied to patients in addition to the routine clinical practice.

Study population will consist of patients with de novo high-aggressive (Gleason 8-10) histologically confirmed mPC diagnosed within 2 years prior to inclusion with available medical history, biopsy formalin-fixed paraffin-embedded (FFPE) tumour tissue sample. It is estimated that approximately 400 patients will be enrolled in about 30 sites.

Demographic and clinical characteristics, treatment approaches and outcomes will be collected during a single visit carried out according to routine clinical practice. Data from the date of de novo high-aggressive mPC diagnosis (date of histological verification) till enrollment will be collected by study physician based on the patient's medical records and interview during the visit and entered into electronic case report form (eCRF). The study physician will be responsible for ensuring that all required data is collected and entered into the eCRF. No follow-up is planned for patients in this study.

For PTEN-loss and HER2-hyperexpression testing (by IHC) and HRRm (mutations in HRR pathway genes), HRD testing (by NGS [next generation sequencing]) available FFPE tumour tissue sample collected as part of routine clinical practice will be used. Testing will be performed in central laboratories.

Overall expected duration of the study enrollment and data collection (from the first patient inclusion to the final database lock) is about 27 months, or until 400 eligible patients are included to the study and data on these patients are collected (including results of FFPE sample testing), whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients aged ≥ 18 years old;
2. Signed ICF, including consent for FFPE tumor tissue sample testing;
3. De novo histologically confirmed high-aggressive (Gleason 8-10) mPC;
4. Diagnosis of mPC (metastatic prostate cancer) within 2 years prior to inclusion;
5. Availability of source medical documentation;
6. Presence of biopsy FFPE tumor tissue sample, obtained as part of standard clinical practice, which will be used for biomarker testing;
7. Unknown HRRm status.

Exclusion Criteria:

1. Participation in any interventional trial since the mPC diagnosis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients aged ≥ 18 years old;
Study Population: It is planned to enroll approximately 400 patients with de novo high-aggressive (Gleason 8-10) histologically confirmed mPC diagnosed within 2 years prior to inclusion in about 30 sites in Russian Federation. Patients must have available medical history and biopsy FFPE tumour tissue sample.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients received any ADT | 24 months
  Proportion of patients received any Androgen deprivation therapy (ADT)
Proportion of patients received ADT by each type and by each drug | 24 months
  Proportion of patients received Androgen deprivation therapy (ADT) by each type and by each drug;
Proportion of patients received first generation antiandrogens | 24 months
  Proportion of patients received first generation antiandrogens;
Proportion of patients received ARPI at mHSPC | 24 months
  Proportion of patients received androgen receptor pathway inhibitors (ARPI) at Metastatic hormone-sensitive prostate cancer (mHSPC) overall and by each drug;
Proportion of patients received any chemotherapy at mHSPC | 24 months
  Proportion of patients received any chemotherapy at Metastatic hormone-sensitive prostate cancer (mHSPC)
Duration of chemotherapy | 24 months
  Duration of chemotherapy in months (to be calculated if chemotherapy completed before or at the enrollment);
Proportion of patients received radiation therapy | 24 months
  Proportion of patients received radiation therapy (RT) overall and by each type (if applicable);
Proportion of patients with each radiation area | 24 months
  Proportion of patients with each radiation area (if applicable) (to be calculated in patients who received any RT);
Proportion of patients underwent surgery at mHSPC stage | 24 months
  Proportion of patients underwent surgery at Metastatic hormone-sensitive prostate cancer (mHSPC) stage overall and by each type (if applicable);
Proportion of patients received triplet therapy | 24 months
  Proportion of patients received triplet therapy (ADT + ARPI + chemotherapy) at mHSPC overall and by each ARPI;
Proportion of patients with PTEN loss by IHC | 24 months
  Proportion of patients with PTEN (Phosphatase and TENsin homolog) loss by Immunohistochemistry (IHC)
Number of Chemotherapy Cycles | 24 months
  Number of chemotherapy cycles is defined as the total number of chemotherapy cycles completed prior to or at the time of study enrollment.

SECONDARY OUTCOMES:
Age at the diagnosis of de novo high-aggressive histologically confirmed mPC | 24 months
  Age at the diagnosis of de novo high-aggressive histologically confirmed mPC, years
Proportion of patients of different races and ethnicities | 24 months
  Proportion of patients of different races and ethnicities
Proportion of patients with presence of a family oncology history | 24 months
  Proportion of patients with presence of a family oncology history (first degree relatives) overall and by each disease;
Proportion of patients with a personal oncology history | 24 months
  Proportion of patients with a personal oncology history overall and by each disease;
Proportion of patients with each category by ECOG assessment | 24 months
  Proportion of patients with each category by ECOG assessment at the inclusion. ECOG is Eastern Cooperative Oncology Group scale used to assess a patient's functional ability (grades are from 0 to 5 where 0 means "Fully active, able to carry on all pre-disease performance without restriction" and 5 means "Dead")
Proportion of patients with each stage by TNM classification | 24 months
  Proportion of patients with each stage by TNM classification. The TNM cancer staging system is a globally recognized method for classifying cancer based on the extent of the tumor (T), involvement of nearby lymph nodes (N), and presence of distant metastasis (M). The TNM values are then grouped into overall stage groupings, usually from I to IV, where Stage I is generally early-stage and Stage IV indicates advanced cancer with distant metastasis.
Proportion of patients with each histological type of tumour | 24 months
  Proportion of patients with each histological type of tumour (types of adenocarcinoma);
Proportion of patients with each category by Gleason scale | 24 months
  Proportion of patients with each category (8 (4+4), 8 (3+5), 8 (5+3), 9, 10)) by Gleason scale. The Gleason scale is a system used to grade prostate cancer based on how different the cancer cells look from normal cells under a microscope. It helps doctors determine how quickly the cancer is likely to grow and spread, influencing treatment decisions. The Gleason score is determined by adding the two most common grades (from 1 to 5) found in the biopsy sample
Proportion of patients with high and low volume of disease | 24 months
  Proportion of patients with high and low volume of disease;
Proportion of patients with each localization of metastases | 24 months
  Proportion of patients with each localization of metastases at the diagnosis, symptomatic or not;
Proportion of patients with each source of tumour sample | 24 months
  Proportion of patients with each source of tumour sample (primary tumour, metastases);
Proportion of patients with each result of HER2 expression by IHC | 24 months
  Proportion of patients with each result of Human Epidermal Growth Factor Receptor 2 (HER2) expression by Immunohistochemistry (IHC). HER2 Status:
  HER2-positive: Cancer cells have high levels of HER2 protein. HER2-negative: Cancer cells have low or no detectable HER2 protein. HER2-low: This category is emerging, indicating a moderate level of HER2 expression, and may be responsive to certain targeted therapies.
Proportion of patients with presence of pathogenic mutations in HRR genes | 24 months
  Proportion of patients with presence of pathogenic mutations in Homologous recombination repair (HRR) genes by Next Generation Sequencing (NGS) results overall and by each gene;
Proportion of patients with positive HRD status | 24 months
  Proportion of patients with positive Homologous recombination deficiency (HRD) status by Next Generation Sequencing (NGS) results.

OTHER OUTCOMES:
Median time from de novo high-aggressive histologically confirmed mPC diagnosis to progression to mCRPC | 24 months
  Median time from de novo high-aggressive histologically confirmed Metastatic prostate cancer (mPC) diagnosis to progression to Metastatic castration-resistant prostate cancer (mCRPC) (calculated between the date of histologically confirmed mPC diagnosis and the date of progression to mCRPC);
Proportion of patients with each site of disease progression | 24 months
  Proportion of patients with each site of disease progression (metastases);
Testosterone level at the time of mCRPC diagnosis | 24 months
  Testosterone level (nmol/l) at the time of castrate-resistant disease (mCRPC diagnosis);
Proportion of low PSA-producing prostate cancer patients at histologically confirmed mPC | 24 months
  Proportion of low PSA-producing prostate cancer patients (PSA <4 ng/ml) at histologically confirmed mPC diagnosis;
Proportion of low PSA-producing prostate cancer patients at progression to mCRPC | 24 months
  Proportion of low PSA-producing prostate cancer patients (PSA <4 ng/ml) at progression to mCRPC;
HRR and HRD concordance | 24 months
  HRR and HRD concordance defined as the proportion of patients with HRD positive or negative status among patients with HRRm (mutations in HRR genes) and HRRwt (wild-type HRR genes).

CONTACTS AND LOCATIONS:
Locations (16):
- Russia (16):
  - Research Site, Arkhangelsk
  - Research Site, Barnaul
  - Research Site, Chelyabinsk
  - Research Site, Irkutsk
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Obninsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
  - Research Site, Saransk
  - Research Site, Tomsk
  - Research Site, Tyumen
  - Research Site, Ufa
  - Research Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Supporting Information: CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/